CLINICAL TRIAL: NCT03835468
Title: The Role of the Microbiota-gut-brain Axis in Brain Development and Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Surrey (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Katherin Cohen-Kadosh, Associate Professor in Developmental Cognitive Neuroscience, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PrebioticExtensionStudyGU2
Record Dates: First submitted 2019-02-01; First posted 2019-02-08 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Gamma-Aminobutyric Acid; Anxiety; Glutamate; Emotion Regulation Abilities
MeSH Terms: conditions — Anxiety Disorders | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two groups. Group 1 will receive a daily dosage of GOS over 4 weeks, whereas group 2 will receive a placebo over the same period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Galacto-oligosaccharides (GOS) Group (Experimental): Participants in this group will receive the daily dosage of galacto-oligosaccharides (GOS) prebiotic for 4 weeks
  Interventions: Dietary Supplement: Galacto-oligosaccharides
- Maltodextrin Group (Placebo Comparator): Participants in this group will receive the daily dosage of Maltodextrin placebo for 4 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharides — GOS is a form of prebiotic, which enhance the growth of beneficial gut bacteria
  Other Names: GOS
  Arms: Galacto-oligosaccharides (GOS) Group
Dietary Supplement: Maltodextrin — sugar based placebo
  Arms: Maltodextrin Group

SUMMARY:
The role of the microbiota-gut-brain axis in brain development and mental health

DETAILED DESCRIPTION:
Anxiety disorders are debilitating conditions that carry enormous individual, social and economic costs. For example, it has been estimated that lifelong persistent mental health problems cost the UK taxpayer £8.6 billion annually. Many mental health problems have their onset in the transitional period from adolescence to early adulthood, possibly a result of the complex and concurrent hormonal, genetic, brain maturational and social changes during this period. Research has shown that brain development and maturation extends well into the third decade of life and that brain activation patterns in late adolescence and early adulthood still differ significantly from mature adults. In the recent years, the microbiome has emerged as a new and important factor that may increase the mental health risk for an individual. The intestine and the brain are intimately connected via the gut-brain axis, which involves bidirectional communication via neural, endocrine and immune pathways. Research in both the human and animal models has also highlighted the important role that intestinal microbiota play in regulating the brain, subsequent behaviour, and particularly in anxiety-like behaviour. Most importantly, it has been shown that the period of adolescence may be a critical window during development where microbiota help fine-tune the gut-brain axis related to stress responses and anxiety.

The research proposed here will investigate the role of the microbiota-gut-brain axis in brain development and mental health. Specifically, the researchers will investigate the effect of prebiotic intake on mental health and well-being in late adolescence/early adulthood, with a particular focus on cortical excitability and connectivity in the emotion regulation brain network.

This research will extend previous research into gut-brain interactions into the final years of adolescence. The period of adolescence is not only important with regards to fine-tuning emotion regulation networks, but also, as has been shown in recent work, critical for establishing healthy gut-brain communication patterns. Specifically, here we will investigate how prebiotic intake (Galacto-oligosaccharides) for 4 weeks affects cognitive functioning, psychological well-being and the underlying brain networks in a sample of 120 female undergraduate students (aged 18-25 years). Specifically, the proposed research has two main aims:

1. To investigate how prebiotic intake affects cortical excitability and plasticity, such as inhibitory GABA/ excitatory glutamate levels in key emotion regulation brain networks.
2. To investigate how prebiotic intake affects psychological functioning and well-being, in particular with regards to anxiety and thought control abilities.

120 participants will be divided into two group of 60 participants, groups will be matched for age, handedness and socio-economic status. At each testing time (Time 1, 2 and 3), participants in both groups will undergo comprehensive behavioural and psychological testing to establish baseline measures of cognitive functioning and psychological well-being (such as anxiety levels).

Each participant will also be asked to collect a stool sample at home for 16s rRNA sequencing of the microbiome at both testing times. Group 1 will receive a daily dosage of GOS over 4 weeks, whereas group 2 will receive a placebo over the same period. In addition, participants from either group will also participate in a brain imaging session to assess the effect of prebiotic supplement intake on the functional responsiveness of emotion regulation brain networks.

For this study, The researchers predict that the intervention group will show improvements in behavioural and psychological variables related to emotion regulation and anxiety in comparison to the placebo group (Hypothesis 1). Predictions also expect to observe decreased excitability in core emotion regulation brain regions such as the amygdala and prefrontal cortex, as assessed via 1H-magnet resonance spectroscopy (Hypothesis 2).

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged between 18-25

Exclusion Criteria:

* Clinical levels of anxiety and/ or co-morbid diagnoses (e.g. depression)
* Current or previous neurological disorders
* Current or previous psychiatric disorders
* Current or previous gastrointestinal disorders
* Current or previous endocrine disorders
* Antibiotic use 3 months prior to the study
* Regular use of pre- and probiotics, including 3 months prior to the study
* Vegan diets

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Changes in brain indices of emotion regulation abilities as a function of prebiotic intake 1 | 4 weeks of intervention
  Increase in brain-based metabolite concentrations (gamma-aminobutyric acid (GABA)) as assessed via Magnetic resonance spectroscopy in the prebiotics group in comparison to the placebo group.
Changes in brain indices of emotion regulation abilities as a function of prebiotic intake 2 | 4 weeks of intervention
  Increase in functional connectivity in brain networks supporting emotion regulation abilities (as assessed via functional magnetic resonance imaging) in the prebiotics group in comparison to the placebo group.
Changes in psychological measures of emotion regulation abilities as a function of prebiotic intake 1 | 4 weeks of intervention
  Decrease in Trait anxiety (State-Trait Anxiety Inventory, Spielberger, 1977) in the prebiotics group in comparison to the placebo group.. For this inventory, a lower overall score is the desired outcome.
Changes in psychological measures of emotion regulation abilities as a function of prebiotic intake 2 | 4 weeks of intervention
  Decrease in Social Anxiety for adolescents (Social Anxiety Scales, La Greca, 1999) in the prebiotics group in comparison to the placebo group. For this scale, a lower overall score is the desired outcome.
Changes in psychological measures of emotion regulation abilities as a function of prebiotic intake 3 | 4 weeks of intervention
  Increase in thought control ability (Thought control ability questionnaire, Luciano et al., 2005) in the prebiotics group in comparison to the placebo group.. For this questionnaire, a higher overall score is the desired outcome.
Changes in gut microbiome composition as a function of prebiotic intake | 4 weeks of intervention
  Increase in beneficial gut bacteria (percentage) in the prebiotics group in comparison to the placebo group. Based on stool sample analyses and microbiome sequencing.
Changes in gut microbiome composition as a function of prebiotic intake | 4 weeks of intervention
  Increase in diversity of gut bacteria in the prebiotics group (number of different bacteria) in comparison to the placebo group. Based on stool sample analyses and microbiome sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Cohen Kadosh, PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No